CLINICAL TRIAL: NCT01802892
Title: An Open Label, Single Center, Adaptive Phase I Study in Healthy Volunteers, to Evaluate the Safety, Efficacy and Dose Responses of SB-751689 (Ronacaleret; a Calcium Sensing Receptor Antagonist)
Brief Title: Study in Healthy Volunteers, to Evaluate the Safety, Efficacy and Dose Responses of SB-751689 (Ronacaleret)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116610
Record Dates: First submitted 2012-11-01; First posted 2013-03-04 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Transplantation, Stem Cell
Keywords: ronacaleret; parathyroid hormone (PTH); CD34+cells; calcium sensing receptor antagonist; hematopoietic stem cells; stem cell mobilization; plerixafor; healthy human volunteer, phase Ib
MeSH Terms: interventions — ronacaleret; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ronacaleret 100 mg (Experimental): Subjects will receive ronacaleret (100 mg once daily) for 5 consecutive days, given in conjunction with a single dose of plerixafor (0.24 mg/kg) SC on the evening of Day 5.
  Interventions: Drug: Ronacaleret 100 mg; Drug: Plerixafor
- Ronacaleret 400 mg (Experimental): Subjects will receive ronacaleret (400 mg once daily) for 5 consecutive days, given in conjunction with a single dose of plerixafor (0.24 mg/kg) SC on the evening of Day 5.
  Interventions: Drug: Ronacaleret 400 mg; Drug: Plerixafor

INTERVENTIONS:
Drug: Ronacaleret 100 mg — Subjects in the Ronacaleret 100 mg group received one tablet orally of ronacaleret 100 mg for 5 consecutive days.
  Arms: Ronacaleret 100 mg
Drug: Ronacaleret 400 mg — Subjects in the Ronacaleret 400 mg group received four tablets orally of ronacaleret 100 mg daily for 5 consecutive days.
  Arms: Ronacaleret 400 mg
Drug: Plerixafor — Subjects in each group received a single dose of plerixafor (0.24mg/kg) SC on the evening of the Day 5 dosing approximately 12 hours before collection of CD34+ cells on day 6.

SUMMARY:
The present study aims to evaluate the impact of 5 days oral administration of ronacaleret 100 miligram (mg) and 400 mg on changes in circulating CD34+ cells, when ronacaleret is followed by the administration of a single dose of plerixafor in healthy human volunteers.

This single centre adaptive design study will be carried out in 2 parts. The part A will evaluate the change in peripheral circulating CD34+ cells in response to two different 5 day regimens of ronacaleret (100 mg or 400 mg once daily), given in conjunction with a single dose of plerixafor (0.24 mg/kilogram [kg]) sub-cutaneously (SC) on the evening of the final days dosing approximately 12 hours before collection of CD34+ cells on day 6. Subjects (5 each) will be assigned to either one of the ronacaleret arms, in an open fashion. Comparisons will be made in the change from baseline to end of treatment peripheral CD34+ cell counts. Part A will be conducted in two cohorts with 5 subjects being enrolled into each of the 2 treatment arms making up the first cohort. Cohort 2 will involve up to 5 further subjects being enrolled into each treatment arm.

The structure of part B will be finalized following a review of data generated in part A.

The total study duration of Part A for each subject including the screening, treatment and follow-up periods will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between 18 and 65 years of age (inclusive).
* Healthy as determined by a physician, based on a medical evaluation and with an estimated Glomerular Filtration Rate (GFR) of >=60 mL/min /1.73 m^2 using the four variable Modification of Diet in Renal Disease (MDRD) equation.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Female of non-child bearing potential, or female subjects and male subjects with female partners of child-bearing potential willing to use protocol-specified methods of contraception to prevent pregnancy during the study.
* Body weight of 55 kg or more and body mass index (BMI) of 20.0 to 35.0 kg/m^2 (inclusive).
* Capable of giving written informed consent.

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive test for HIV, B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of or therapy for osteoporosis
* Subject has had treatment for any condition relating to the thyroid/parathyroid gland which in the opinion of the investigator may influence the subjects production of PTH
* Subjects with any contraindications or know allergies to receiving plerixafor
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones).
* Subjects taking calcium and/or vitamin D supplements, during or within 2 weeks of study initiation
* Subjects taking any concomitant medications
* Specific laboratory abnormalities at screening like Serum calcium (total or albumin-adjusted) outside the central laboratory reference range, PTH outside the normal range, Creatine phosphokinase (CPK) outside the normal range
* Subjects with abnormal Vitamin D (Vitamin D, 25-Hydroxy) levels may be enroled if repeat lab results, obtained within 14 days of initial screening assessments, are within the normal range
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females.
* Lactating or pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* The subject has participated in a clinical trial within 30 days or 5 half-lives of the IP prior to the first dosing day in the current study.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2013-04-02 (Actual); Study Completion 2013-04-02 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in CD34+ cell counts | Baseline and upto Day 14
  The mean fold change from baseline in the number of circulating CD34+ cells for all treatment arms will be assessed. Samples will be collected at screening, Day 4 and Day 5 (2 hrs post ronacaleret dose), Day 6 (12 hrs and 14 and 16 hrs post plerixafor dose) and Day 14

SECONDARY OUTCOMES:
Spontaneous AE reporting | Up to 14 days
  Adverse events (AEs) will be collected from the start of Investigation Product (IP) and until the follow-up visit
Clinical laboratory safety data | Up to 14 days
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis
Measure of vital signs to access safety and tolerability | Up to 14 days
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate. Subjects should have been in a supine or semi-supine (recumbent) position for at least 5 minutes prior to taking measurements
PTH responses | Up to 6 days
  Parathyroid hormone (PTH) has been shown to stimulate osteoblasts and osteoclasts and also associated with increased numbers of circulating CD34+ve cells
Quantification of the number of stem cells | Part B will be detailed in an amendment to the protocol following a data review of part A
  The number of stem cells from the various hematopoietic lineages through colony forming unit assays in Part B of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Results for study 116610 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116610?search=study&study_ids=116610#rs